CLINICAL TRIAL: NCT02079714
Title: Streamlining Trauma Research Evaluation With Advanced Measurement: STREAM Study
Brief Title: Streamlining Trauma Research Evaluation With Advanced Measurement
Acronym: STREAM
Status: Completed | Type: Observational
Sponsor: Major Extremity Trauma Research Consortium (Other)
Responsible Party: Sponsor
Other Study IDs: 1R01AR064066-01 (NIH)
Record Dates: First submitted 2014-02-24; First posted 2014-03-06 (Estimated); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Orthopaedic Trauma
Keywords: Orthopaedic Trauma; Injury
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Questionnaire: All STREAM Study participants will be complete a series of computer adaptive testing (CAT) questions covering all core and exploratory domains, once written informed consent is obtained. Administration of these surveys will follow completion of all other follow-up activities related to the main METRC study in which they were originally enrolled. Identical surveys will be repeated at the 6 month study visit. At the final 12 month study visit, participants will complete the CAT survey for the six core domains, and will also complete a randomly assigned subset of items from the total item bank across these six core domains. At any visit, if the CAT cannot be administered, respondents will instead complete paper surveys of the short form for each domain.

SUMMARY:
The STREAM Study is a prospective longitudinal observational outcomes study that will examine the reliability, validity and responsiveness of the PROMIS tools for clinical research following orthopaedic trauma.

DETAILED DESCRIPTION:
Objective: As part of the NIH Roadmap initiative, PROMIS (patient reported outcomes measurement information system) has developed tools, including item banks, short forms and computer-adaptive tests (CATs) that can help standardize measurement for many health-related quality of life domains. These PROMIS tools are being tested in large general population samples across the lifespan. The overall goal of the present study is to assess the performance and research utility of these new tools in new patient populations for future comparative effectiveness research projects. The proposed project will examine the reliability, validity and responsiveness of the PROMIS tools for clinical research following orthopaedic trauma.

Specific Aim 1: Examine the measurement properties of existing PROMIS CATs and item banks in patients with orthopaedic trauma. Investigators will incorporate ten (six core and four exploratory) PROMIS short form and CATs into the longitudinal data collection of five ongoing orthopaedic trauma clinical trials and administer an expanded data collection interview at the time of their last study follow up which will be used to:

1a: Evaluate reliability and construct validity of the PROMIS CATs

1b: Compare measurement precision of the six existing item banks when applied in an orthopaedic trauma population versus the general population.

1. c: Identify items from existing PROMIS item banks that function differently in our population compared with the general population.

   Specific Aim 2: Examine the responsiveness of existing PROMIS domains in patients with orthopaedic trauma. Specifically, investigators will:
2. a: Examine the responsiveness of PROMIS domains against expected clinical recovery in this population.

2b: Examine the responsiveness of PROMIS domains against well-defined clinical inflection points in the recovery process, such as infections, non-unions, flap failures, and other complications.

2c: Examine the responsiveness of PROMIS domains against treatment effects observed for interventions being studied in these trials, which include a psychosocial intervention, a pharmacologic intervention, and a device. These trials are being evaluated using widely used traditional outcome measurement tools.

Specific Aim 3: Study the integration of the PROMIS tools within the data collection infrastructure of METRC. Key feasibility components examined will be integration with our distributed electronic data capture system (REDCap), and use of the CAT technology across dozens of trauma centers and orthopaedic trauma clinics.

3a. Compare the rate of use of CAT-based assessment versus short-form data collection 3b: Compare the data completeness using existing METRC approaches, CAT and short form PROMIS instruments 3c: Compare respondent burden using existing METRC approaches, CAT and short form PROMIS instruments.

Study design: The STREAM study is a multi-center, prospective longitudinal observational study to evaluate the reliability, validity and responsiveness of PROMIS tools in orthopaedic trauma patients.

ELIGIBILITY:
Any patient participating in the FIXIT, OUTLET, TAOS, OXYGEN, VANCO or Pain studies returning for a 3 month follow-up visit is eligible for participation in the proposed STREAM study. Respondents who are unable to give informed consent (or would require a proxy) at the time of the 3 month visit will be excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Orthopaedic trauma patients who are currently enrolled in the PAIN, FIXIT, OUTLET, OXYGEN, VANCO or TAOS METRC studies. These studies look at outcomes following injuries to the foot, ankle, tibia etc.
Sampling Method: Probability Sample
Enrollment: 1065 (Actual)
Dates: Start 2014-01; Primary Completion 2019-06 (Actual); Study Completion 2020-10 (Actual)

PRIMARY OUTCOMES:
Reliability and Validity | 9 months
  The primary endpoint for this study is the reliability and construct validity of the PROMIS CAT instruments.

SECONDARY OUTCOMES:
Responsiveness | 9 months
  Responsiveness against clinical recovery, inflection points and effective interventions.
Data Completion | 9 months
  Data completeness in CAT-based instruments vs short form paper-based data collection
Participant Burden | 9 months
  Respondent burden, as indicated by time to complete instrument, which will be recorded by the CAT, and manually recorded at start/stop time on the paper short forms

CONTACTS AND LOCATIONS:
Locations (44):
- United States (44):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Naval Medical Center San Diego, San Diego, California
  - University of California San Francisco Medical Center, San Francisco, California
  - Denver Health and Hospital Authority, Denver, Colorado
  - University of Miami Ryder Trauma Center, Miami, Florida
  - Orlando Regional Medical Center, Orlando, Florida
  - Tampa General Hospital, Tampa, Florida
  - Orthoindy at St Vincent, Indianapolis, Indiana
  - Eskenazi Hospital, Indianapolis, Indiana
  - OrthoIndy / Methodist Hospital, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - Louisiana State University, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center, Shreveport, Louisiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Orthopaedic Associates of Michigan, Spectrum Health, Grand Rapids, Michigan
  - Hennepin County Medical Center / Regions Hospital, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Barnes Jewish Hospital, St Louis, Missouri
  - St. Louis Medical Center, St Louis, Missouri
  - Jamaica Hospital Medical Center, Jamaica, New York
  - Mission Hospital, Asheville, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Duke University Hospital, Durham, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - MetroHealth Medical Center, Cleveland, Ohio
  - Grant Medical Center, Columbus, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Geisinger Health System, Danville, Pennsylvania
  - Penn State University M.S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - York Hospital, York, Pennsylvania
  - Rhode Island Hospital, Brown University, Providence, Rhode Island
  - Vanderbilt Medical Center, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - San Antonio Miliary Medical Center, Fort Sam Houston, Texas
  - University of Texas Health Science Center - Houston, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
  - Naval Medical Center Portsmouth, Portsmouth, Virginia
  - University of Washington Harborview, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin